CLINICAL TRIAL: NCT05984849
Title: A Pilot Randomized Controlled Study to Examine Feasibility and Preliminary Effectiveness of a Game-based Intervention in Promoting HPV Vaccination Among Vulnerable Youth to Prevent Cancers
Brief Title: Playing Game to Learn About Children's Vaccine Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Angela Chia-Chen Chen, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FP00033005
Record Dates: First submitted 2023-07-25; First posted 2023-08-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: HPV; Vaccine-Preventable Diseases
Keywords: adolescent; game intervention
MeSH Terms: conditions — Vaccine-Preventable Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV game group (Experimental): parent-child dyads receive HPV game intervention
  Interventions: Behavioral: vaccination game
- Usual care (No Intervention): parent-child dyads receive usual care (no intervention)

INTERVENTIONS:
Behavioral: vaccination game — A health game to promote HPV vaccination among youth
  Arms: HPV game group

SUMMARY:
This proposed study aims to conduct timely research that promotes vaccine confidence and vaccination of one strongly recommended vaccine with suboptimal uptake rates: Human papillomavirus (HPV) in vulnerable and underserved youth aged 11-14.

DETAILED DESCRIPTION:
The study objectives are:

Objective 1: Assess feasibility (participation rate, retention, involvement, satisfaction) of one game-based interventions targeting HPV vaccination.

Objective 2: Conduct a pilot RCT with three conditions (Arm 1: HPV game-based intervention; Arm 2: usual care). The investigators will explore patterns of pre- to post-intervention change in theoretical mediators and vaccine intent, and explore levels of vaccine intent and uptake in 90 parent-child dyads of unvaccinated youth aged 11-14.

ELIGIBILITY:
Inclusion Criteria:

* Child sample: (1) 11-14 years old, (2) speaks and reads English, (3) has never received any doses of the HPV vaccine, (4) is not currently enrolled in another project that involves HPV-related education, and (5) agrees and provides assent to participate in research activities.
* Parent sample: (1) parent or legal guardian of the participating child, (2) speak and read English, (3) own a smartphone, (4) agree to receive email and text messages, (5) is not currently enrolled in another project that involves HPV-related education, and (6) agree and provide consent to participate in research activities.

Exclusion Criteria: Individuals who do not meet inclusion criteria or refuse to provide consent/assent.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of eligible individuals agreeing to participate | T0 (occurs after consenting and before assigning to different study conditions)
  Assessed by the % of eligible individuals agreeing to participate
Proportion of participants who are retained through follow-up | T2 (occurs two months after completion of the intervention)
  Assessed by the % of participants who are retained through follow-up
Percentage of participants who complete the intervention and assessments | T2 (occurs two months after completion of the intervention)
  Assessed by the % of participants who complete the intervention and assessments
Participant satisfaction with the project | T2 (occurs two months after completion of the intervention)
  Assessed by two Likert scale questions: (1) are you satisfied with the program? (2) Will you recommend this program to others? Responses: from (1) very dissatisfied/definitely not to (5) very satisfied/definitely yes)
Intention to vaccinate the children against HPV | T0 (occurs after consenting and before assigning to different study conditions); T1 (occurs immediately post intervention);T2 (occurs two months after completion of the intervention)
  Assessed by a Likert scale question: How likely will you (parent) vaccinate your child against HPV? Responses: (0) no; (1) maybe; (2) yes

SECONDARY OUTCOMES:
Children receives the first dose of HPV vaccine | T2 (occurs two months after completion of the intervention)
  Assessed by one binary question regarding whether or not the child has received the first dose of HPV vaccine. Responses: yes, no

CONTACTS AND LOCATIONS:
Overall Officials: ANGELA C CHEN, PhD, Principal Investigator — Michigan State University
Locations (1):
- Community, Chandler, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, non-sensitive data will be deposited in Dryad no later than the date of publication.
Time Frame: Start: no later than the date of publication End: remain publicly available for 3 years following publication
Access Criteria: All users will have open access to the data without restriction, consistent with Dryad's open-access model. Data can be accessed directly through Dryad's website using the assigned DOI, ensuring discoverability and persistent availability. No personally identifiable or sensitive information will be shared.